CLINICAL TRIAL: NCT05518682
Title: Assessment of Bimodal Stimulation Device Compliance and Satisfaction in Individuals With Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Neuromod Devices Limited (Unknown); Kent Taylor (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00015524
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: One arm with the same device protocol, except that there are two subgroups with different hearing/audiogram profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single study arm (Experimental): The Lenire device is CE marked in Europe and intended to reduce the symptoms of tinnitus. It comprises a handheld controller and an intra-oral device called a Tonguetip® Intra-Oral Device (IOD), which delivers gentle electrical stimulation to the tongue, and also comprises of a set of wireless consumer headphones that deliver audio stimulation. The sound and tongue stimulus parameters such as stimulus rate, stimulus intensity, and the timing relationship between the auditory and somatosensory stimulus events are grouped into stimulation Parameter Sets (PS). PS1 is used during the first 6-weeks of stimulation and PS4 is used during the second 6-weeks of stimulation, similar to what is routinely used for tinnitus individuals in Europe. For this study, the device software has been modified to allow users to adjust the headphone volume to a level that is comfortable and clearly audible instead of a preset volume with limited adjustments based on the patient's audiogram.
  Interventions: Device: Lenire bimodal stimulation device

INTERVENTIONS:
Device: Lenire bimodal stimulation device — The sound and tongue stimulus parameters such as stimulus rate, stimulus intensity, and the timing relationship between the auditory and somatosensory stimulus events are grouped into stimulation Parameter Sets (PS). PS1 is used during the first 6-weeks of stimulation and PS4 is used during the second 6-weeks of stimulation, similar to what is routinely used for tinnitus individuals in Europe.
  Other Names: PS1-PS4

SUMMARY:
The research objective of the proposed usability study is to assess the compliance and acceptance/satisfaction of using a bimodal stimulation device with the ability to self-adjust the sound stimulus presented to the ears via headphones. In particular, the CE marked bimodal stimulation portable device, Lenire, which is developed by Neuromod Devices Limited (Dublin, Ireland) to alleviate the symptoms of chronic subjective tinnitus, is currently configured according to a tinnitus person's audiogram (i.e., hearing threshold profile for different sound frequencies) during fitting in a hearing center. Lenire device is a non-invasive stimulation device that consists of a controller that connects to headphones for sound delivery to the ears and connects to a mouth component that provides gentle electrical stimulation to the tongue surface. Individuals are recommended to use the device for 60 minutes daily (two 30-minute sessions consecutively or at different times of the day) for at least 10 weeks. Lenire is already commercialized across Europe and available by audiologists or hearing technicians in numerous hearing centers for treating tinnitus. It has also been evaluated in two large-scale clinical trials in over 500 tinnitus participants, demonstrating tinnitus benefit and minimal risk with high compliance and satisfaction rates.

The primary objective of the proposed usability study is to first assess compliance and satisfaction with the Lenire device that does not require an audiogram for fitting and that can be implemented mostly through virtual visits (except for the first visit). These modifications to the Lenire fitting process will reduce the time and personnel effort required for its implementation, enabling a broader patient population to access bimodal stimulation for tinnitus treatment, including military personnel and those who are not nearby hearing centers for in-person sessions. High compliance and satisfaction rates from this small proof-of concept usability study will then justify and guide a larger clinical study to assess efficacy and performance of this newly implemented Lenire device process.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over at time of consent
* Ability to read and understand English
* Willing and able to provide and understand informed consent
* Willing to commit to the full duration of the investigation
* Subjective tinnitus
* Tinnitus duration of greater than or equal to 3 months and less than or equal to 20 years at time of consent
* Baseline THI score from 38 to 76
* Hearing loss condition (low hearing loss group (n=10) and high hearing loss group (n=10))
* Access to reliable internet connection and device to complete virtual video visits and electronic surveys

Exclusion Criteria:

* Subjective tinnitus, where pulsatility is the dominant feature
* Objective tinnitus
* Middle ear pathology in either ear including documented/known conductive hearing loss >= 20 dB at three adjacent frequencies or if a diagnosis of a tympanic membrane perforation or other middle ear pathology has been rendered, if there is an indwelling pressure equalization tube by patient report, or if middle ear surgery has been performed
* Began wearing hearing aids within the past 3 months
* Health care provider has rendered a diagnosis of Meniere's disease or other disorder with fluctuating hearing loss
* A diagnosis of hyperacusis, misophonia or hypersensitivity to loud noises has been rendered
* History of auditory hallucinations
* Tumor on the hearing or balance nervous systems
* Hospitalization, or visit to a physician, for a head or neck injury, including whiplash, in the previous 12 months
* Initiated new prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics. See Appendix 2 for list of medical treatments.
* Ceased prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics. See Appendix 2 for list of medical treatments.
* Changed dosage of prescription medications in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics. See Appendix 2 for list of medical treatments.
* Any use of benzodiazepines or sedative hypnotics (either regularly or on demand)
* Neurological condition that may lead to seizures or loss of consciousness (e.g., epilepsy)
* Participant with a pacemaker or other electro-active implanted device
* Participant previously diagnosed with psychosis or schizophrenia
* Participants diagnosed with Burning Mouth Syndrome
* A diagnosis of bothersome temporomandibular joint disorder (TMJ) has been rendered
* Previous involvement in a clinical investigation for tinnitus treatment or had an implantable or surgical intervention for tinnitus
* Inability to physically or comprehensively use the device
* Oral piercings that cannot or will not be removed
* Current or previous involvement in medico-legal cases
* Pregnancy per patient report
* Prisoner
* PI does not deem the candidate to be suitable for the investigation for other reasons not listed above. Rationale must be provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2025-02-16 (Actual)

PRIMARY OUTCOMES:
Compliance rate after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation)
  Compliance rate after 12 weeks of bimodal stimulation with minimum compliance of a total of 36 hours

SECONDARY OUTCOMES:
Satisfaction rate after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation)
  Satisfaction rate (two satisfaction questions) after 12 weeks of bimodal stimulation

OTHER OUTCOMES:
Impact of the stimulation device on tinnitus symptoms after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation) and 12 week follow-up visit
  Tinnitus Handicap Inventory (THI)
Impact of the stimulation device on tinnitus symptoms after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation) and 12 week follow-up visit
  Tinnitus Functional Index (TFI)
Impact of the stimulation device on tinnitus symptoms after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation) and 12 week follow-up visit
  Visual Analog Scale for Loudness (VAS-L)
Impact of the stimulation device on health after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation)
  Patient Health Questionnaire (PHQ-8)
Impact of the stimulation device on stress after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation)
  Perceived Stress Scale (PSS-10)
Impact of the stimulation device on anxiety after 12 weeks of bimodal stimulation | Enrollment visit to week 12 visit (end of device stimulation)
  Generalized Anxiety Disorder (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Adams, MD, Principal Investigator — University of Minnesota; Peggy Nelson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - TESSLab/PWB, Minneapolis, Minnesota, United States